CLINICAL TRIAL: NCT02213770
Title: Long Term Effect of High-intensity Training After Heart Transplantation
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Health Association (Other)
Responsible Party: Principal Investigator, Marianne Yardley, Cand med, Oslo University Hospital
Other Study IDs: 2014/872/REK sør-øst C
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Heart Transplant Recipients

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blodsamples from the patients will be studied:
  Standard samples: RBC, WBC, plates, CRP, kreatinin, urea, liver tests, thyorid gland tests, lipid profile, fasting- glucose og hba1c, Pro BNP, troponin T, uric acid.
  Supplement: Inflammation cytokines/chemokines such as TNF alfa, sTNFR2 og IL-6, IL-10, MCP-1 og IL-8. Growth factors and inhibitors for innervation. Markers for endothelial function; endotelin and von- Willebrand faktor and anti- trombotic factors; fibrinogen, plasminogen activator inhibitor-1.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention group: Group that followed high- intensity interval training program in TEX study.
- Control group: Followed up on a regular basis for HTx recipients in Norway.

SUMMARY:
High-intensity training (HIT) has repeatedly been documented to have superior positive effects compared to moderate exercise in patients with coronary heart disease and heart failure. Since heart transplant recipients (HTx), have a denervated heart with different respond to exercise, HIT has previously not been introduced among these patients. Rikshospitalet carried out a RCT to investigate this (the TEX study 2009-2012), and found that this form of exercise also was highly effective and safe in long term HTx with clinically significant improvement in VO2peak, muscular exercise capasity, general HRQoL, and even slower progression of CAV (coronary allograft vasculopathy). Based on these findings we ask the following questions in this follow-up study:

1. Would the effect on VO2peak, HRQoL,muscle capacity and CAV obtained during the study period continue during long term follow up (5 years)?
2. Is the intervention group more physical active after HIT compared to the control group?

ELIGIBILITY:
Inclusion Criteria:

* stable situation
* optimal medical treatment
* written concent

Exclusion Criteria:

* unstable situation,
* infections (open wounds or skin diseases),
* physical conditions that prevents participation,
* or other injuries/ diseases who are contraindicated with training.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The TEX population.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
mean VO2peak in the intervention group and control group | 5 years after start of inclusion in RCT (TEX). One measurment.
  We will use the same test protocol as the TEX- study.

SECONDARY OUTCOMES:
How many has progression of cardiac allograft vasculopathy in the intervention group and control group. | 5 years after inclusion in RCT (TEX study).
  Progression of vasculopathy will be studied with IVUS technique, and compared with IVUS pictures from TEX.
Mean muscle capacity in the intervention group and control group. | 5 years after inclusion in RCT, TEX study.
Quality of life | 5 years after inclusion in TEX- study.
  We will use validated questionnaires to estimate quality of life and to evaluate depression.
Difference in activity level between groups | 5 years after inclusion i RCT, TEX study.
  To estimate activity the study population will fill out a validated questionnaire about physical activity, and they will wear a physical activity monitor at home for one week.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Gullestad, professor, Study Director — OUS- kardiologisk avdeling
Locations (1):
- OUS- Rikshospitalet, Oslo, Oslo County, Norway

REFERENCES:
- [Result] Nytroen K, Myers J, Chan KN, Geiran OR, Gullestad L. Chronotropic responses to exercise in heart transplant recipients: 1-yr follow-up. Am J Phys Med Rehabil. 2011 Jul;90(7):579-88. doi: 10.1097/PHM.0b013e31821f711d. PMID 21765276
- [Result] Nytroen K, Rustad LA, Gude E, Hallen J, Fiane AE, Rolid K, Holm I, Aakhus S, Gullestad L. Muscular exercise capacity and body fat predict VO(2peak) in heart transplant recipients. Eur J Prev Cardiol. 2014 Jan;21(1):21-9. doi: 10.1177/2047487312450540. Epub 2012 Jun 1. PMID 22659939
- [Result] Nytroen K, Rustad LA, Erikstad I, Aukrust P, Ueland T, Lekva T, Gude E, Wilhelmsen N, Hervold A, Aakhus S, Gullestad L, Arora S. Effect of high-intensity interval training on progression of cardiac allograft vasculopathy. J Heart Lung Transplant. 2013 Nov;32(11):1073-80. doi: 10.1016/j.healun.2013.06.023. Epub 2013 Jul 29. PMID 23906899
- [Result] Nytroen K, Rustad LA, Aukrust P, Ueland T, Hallen J, Holm I, Rolid K, Lekva T, Fiane AE, Amlie JP, Aakhus S, Gullestad L. High-intensity interval training improves peak oxygen uptake and muscular exercise capacity in heart transplant recipients. Am J Transplant. 2012 Nov;12(11):3134-42. doi: 10.1111/j.1600-6143.2012.04221.x. Epub 2012 Aug 17. PMID 22900793